CLINICAL TRIAL: NCT07395778
Title: Nasojejunal Feeding Versus Oral Feeding Following Endoscopic Drainage of Walled Off Pancreatic Necrosis: A Randomized Controlled Pilot Study
Brief Title: Nasojejunal Feeding Versus Oral Feeding Following Endoscopic Drainage of Walled Off Pancreatic Necrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Saurabh Kumar Singh, Senior Resident, Department of Gastroenterology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IEC-INT/2025/DM-3119
Record Dates: First submitted 2025-11-18; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Walled Off Pancreatic Necrosis; Acute Pancreatitis (AP); Endoscopic Ultrasound-Guided Drainage
Keywords: Cystogastrostomy, Walled off pancreatic necrosis, nutrition
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasojejunal feeding arm (Experimental)
  Interventions: Procedure: endoscopic ultrasonography guided cystogastrostomy
- Oral feeding (Active Comparator)
  Interventions: Procedure: endoscopic ultrasonography guided cystogastrostomy

INTERVENTIONS:
Procedure: endoscopic ultrasonography guided cystogastrostomy — Nasojejunal tube will be placed post EUS-CG or oral diet would be started after randomization

SUMMARY:
The goal of this randomized control trial is to assess whether nasojejunal feed is better than oral nutrition in patients who are undergoing endoscopic cystogastrostomy of walled off necrosis following acute pancreatitis. It will also try to answer, the incidence of infections and feed tolerance.

The main question it tries to answer is

1. whether nasojejunl feed is better than oral feed in patients undergoing endoscopic cystogastrostomy in walled off necrosis following acute pancreatitis
2. How much infections they develop, whether they are able to tolerate the feed, weight gain and reintervention rates in each group

ELIGIBILITY:
Inclusion Criteria:

1. Patients of acute pancreatitis (AP) with 18-75 years of age
2. Patients with symptomatic WON requiring EUS guided transluminal drainage
3. Provision of written informed consent

Exclusion Criteria:

1. Patients with collection not amenable for EUS guided drainage (distance of WON >1 cm from the gastrointestinal lumen)
2. Known malignancy or immunocompromised state
3. Previous upper gastrointestinal(GI) surgery interfering with absorption
4. Active GI bleeding
5. GI obstruction, ileus or persistent vomiting
6. Patients moribund to undergo endoscopic procedure (Glasgow coma scale <8 or patients on ventilatory support)
7. Patients with irreversible coagulopathy like platelets <50,000/mm3 and/or INR>1.5
8. Pregnant or lactating female

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Nutritional failure | 14 days
  To compare the rate of nutritional failure at Day 14 between Nasojejunal and oral feeding post endoscopic transmural drainage of WON

SECONDARY OUTCOMES:
Infection and new onset organ failure | 14 days
  To compare infection rates, need for antibiotic escalation and new onset organ failure
Re-intervention needs | 14 days
  To compare the need for re-intervention and hospital stay duration in either of the group
Change in weight | 14 days
  To compare patient weight
Inflammatory markers | 14 days
  To compare change in inflammatory markers (CRP, Serum Albumin)

CONTACTS AND LOCATIONS:
Overall Officials: Surender Singh Rana, Professor, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After 1 year
Access Criteria: Who wants to publish individual data meta-analysis

DOCUMENTS (2):
  • Study Protocol: Study Protocol (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT07395778/Prot_000.pdf
  • Informed Consent Form (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT07395778/ICF_001.pdf